CLINICAL TRIAL: NCT00374205
Title: A Comparative Assessment of the Effectiveness of Artemether Plus Lumefantrine Versus Artesunate Plus Amodiaquine for the Treatment of Children With Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Randomized Trial on Effectiveness of ACTs in Ghana
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim analysis showed more LCFs in one of the treatment arms
Sponsor: Bernhard Nocht Institute for Tropical Medicine (Other Government)
Collaborators: Presbyterian Health Service (PHS) (Unknown); Kumasi Centre for Collaborative Research (KCCR) (Other); School of Medical Sciences Kumasi (SMS/KNUST) (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01KA22062006
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Malaria, Falciparum
Keywords: Ghana; Effectiveness; Safety; Drug-Resistance; ACT; Coartem; Arsucam
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artesunate; Amodiaquine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AL (Experimental): Artemether plus Lumefantrine 6 dose 3 days treatment
  Interventions: Drug: Artemether-Lumefantrine
- ASAQ (Active Comparator): Artesunate plus Amodiaquine
  Interventions: Drug: Artesunate plus Amodiaquine

INTERVENTIONS:
Drug: Artesunate plus Amodiaquine — Artesunate 50 mg and Amodiaquine 153 mg co-blister tablets: 3 days once daily weight-adjusted dosing according to manufacturer
  Other Names: Arsucam®
  Arms: ASAQ
Drug: Artemether-Lumefantrine — Artemether 20 mg/Lumefantrine 120mg fixe-dose-combination tablets: 3 days twice daily weight-adjusted dosing according to manufacturer
  Other Names: Coartem®
  Arms: AL

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of two Artemisinin Combination Therapies (ACTs) for the treatment of children with uncomplicated Plasmodium falciparum malaria

DETAILED DESCRIPTION:
Childhood mortality related to Plasmodium falciparum malaria is on the rise with more than 1 million deaths per year in Sub-Saharan Africa. In the context of growing drug-resistance to antimalarials health officials are calling for rapid replacement of failing drugs by combining antimalarial drugs. Artemisinin Combination Antimalarial Therapies (ACTs) are in the focus of malaria control programmes and are recommended for first-line treatment in African countries. ACTs have been reported to be highly effective as artemisinin derivatives cause a rapid and substantial decrease in the parasite load when used for treating patients with malaria and resistance to artemisinin is still lacking. However, the short half-lives of artemisinins result in frequent recrudescent infections when used alone and therefore, much interest lays on the choice of the combination partner drug. ACTs also have been proposed as a means of reducing transmission by the reduction of gametocytes and of delaying the spread of drug resistance and prolonging the therapeutic life span of. Nevertheless, drug resistance of parasites to the respective partner drug is a matter of concern. Artesunate-amodiaquine (AQ) and artemether-lumefantrine (AL) are two registered fixed-dose artemisinin combination chemotherapies used in Africa which are GMP-manufactured at industrial scale. There is still limited data from randomised, controlled trials to support the general effectiveness of these two ACTs in Africa, including Ghana. More data is needed to compare these two therapies to make evidence-based first-line treatment decisions. Importantly, it is difficult to predict how combination therapy may affect the spread of drug resistance and monitoring drug resistance markers should be embedded in these trials to guide drug policy decision.

The aim of this open-labelled, randomised drug trial is to compare the effectiveness and safety of artesunate-amodiaquine (Arsucam®) against artemether plus lumefantrine (Coartem®) for the treatment of children under five years of age with uncomplicated Plasmodium falciparum malaria.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients aged 6 months to 59 months
* Absence of severe malnutrition
* A slide-confirmed P. falciparum asexual parasitaemia between 2,000/µl and 200,000/µl
* A measured axillary temperature ≥ 37.5 °C or rectal/tympanic temperature ≥ 38.0 °C
* Absence of general danger signs (unable to drink; repeated vomiting; recent history of convulsions; lethargic or unconscious state; unable to stand up or to sit)
* Ability to tolerate oral therapy
* Permanent residence in study area
* Informed consent by the legal representative of the subject, if possible, the parents

Exclusion Criteria:

* Adequate anti-malarial treatment within the previous 7 days
* Antibiotic treatment for a current infection
* Previous participation in a clinical trial
* Haemoglobin < 5 g/dl
* Leucocyte count: > 15000/µl
* Mixed plasmodial infection
* Severe malaria as defined by WHO recommendations
* Any other severe underlying disease (cardiac, renal, hepatic diseases, malnutrition, known HIV infection) or concomitant disease masking assessment of response
* History of allergy or intolerance against trial medication

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 245 (Actual)
Dates: Start 2006-09; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Clinical and PCR-controlled parasitological cure rate at day 28 | 28 days

SECONDARY OUTCOMES:
Clinical and PCR-controlled parasitological cure rate at day 14 | 14 days
Effect on anaemia | 28 days
Molecular Drug Resistance Markers | 28 days
Recrudescence and Reinfection | 28 days
Effects on Gametocytemia | 28 days
Acceptance of Therapies | 7 days
Incidences of malaria episodes over a follow-up period of 1 year | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ansong, MD, Principal Investigator — School of Medical Science (SMS), Kwame Nkrumah University of Science and Technology (KNUST), Kumasi, Ghana
Locations (1):
- Agogo Presbyterian Hospital, Agogo, Asante Akim North District, Ghana

REFERENCES:
- [Background] Bukirwa H, Yeka A, Kamya MR, Talisuna A, Banek K, Bakyaita N, Rwakimari JB, Rosenthal PJ, Wabwire-Mangen F, Dorsey G, Staedke SG. Artemisinin combination therapies for treatment of uncomplicated malaria in Uganda. PLoS Clin Trials. 2006 May;1(1):e7. doi: 10.1371/journal.pctr.0010007. Epub 2006 May 19. PMID 16871329
- [Background] Mutabingwa TK, Anthony D, Heller A, Hallett R, Ahmed J, Drakeley C, Greenwood BM, Whitty CJ. Amodiaquine alone, amodiaquine+sulfadoxine-pyrimethamine, amodiaquine+artesunate, and artemether-lumefantrine for outpatient treatment of malaria in Tanzanian children: a four-arm randomised effectiveness trial. Lancet. 2005 Apr 23-29;365(9469):1474-80. doi: 10.1016/S0140-6736(05)66417-3. PMID 15850631
- [Background] Makanga M, Premji Z, Falade C, Karbwang J, Mueller EA, Andriano K, Hunt P, De Palacios PI. Efficacy and safety of the six-dose regimen of artemether-lumefantrine in pediatrics with uncomplicated Plasmodium falciparum malaria: a pooled analysis of individual patient data. Am J Trop Med Hyg. 2006 Jun;74(6):991-8. PMID 16760509
- [Background] Price RN, Uhlemann AC, van Vugt M, Brockman A, Hutagalung R, Nair S, Nash D, Singhasivanon P, Anderson TJ, Krishna S, White NJ, Nosten F. Molecular and pharmacological determinants of the therapeutic response to artemether-lumefantrine in multidrug-resistant Plasmodium falciparum malaria. Clin Infect Dis. 2006 Jun 1;42(11):1570-7. doi: 10.1086/503423. Epub 2006 Apr 26. PMID 16652314
- [Background] Martensson A, Stromberg J, Sisowath C, Msellem MI, Gil JP, Montgomery SM, Olliaro P, Ali AS, Bjorkman A. Efficacy of artesunate plus amodiaquine versus that of artemether-lumefantrine for the treatment of uncomplicated childhood Plasmodium falciparum malaria in Zanzibar, Tanzania. Clin Infect Dis. 2005 Oct 15;41(8):1079-86. doi: 10.1086/444460. Epub 2005 Sep 13. PMID 16163624
- [Background] Sidhu AB, Uhlemann AC, Valderramos SG, Valderramos JC, Krishna S, Fidock DA. Decreasing pfmdr1 copy number in plasmodium falciparum malaria heightens susceptibility to mefloquine, lumefantrine, halofantrine, quinine, and artemisinin. J Infect Dis. 2006 Aug 15;194(4):528-35. doi: 10.1086/507115. Epub 2006 Jul 11. PMID 16845638
- See also: Homepage of the Kumasi Centre for Collaborative Research (study site) — http://www.kccr.de/kccr/